CLINICAL TRIAL: NCT03383679
Title: A Randomized Phase 2 Study in Patients With Triple-negative Androgen Receptor Positive Locally Recurrent (Unresectable) or Metastatic Breast Cancer Treated With Darolutamide or Capecitabine
Brief Title: Study on Androgen Receptor and Triple Negative Breast Cancer
Acronym: START
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UNICANCER (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UC-0140/1711 - UCBG3-06; 2017-002284-18 (EudraCT Number)
Record Dates: First submitted 2017-10-13; First posted 2017-12-26 (Actual); Last update posted 2022-11-21 (Actual); Status verified 2022-11

CONDITIONS: Breast Cancer Female; Triple Negative and Androgen Receptor Positive
MeSH Terms: interventions — darolutamide; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 Darolutamide (Experimental): Darolutamib: 600 mg (2 tablets of 300 mg) twice daily with food (equivalent to a daily dose of 1200 mg) will be administered orally, continuously until disease progression
  Interventions: Drug: Darolutamide
- Arm 2 Capecitabine (Other): according to the 3rd ESO-ESMO international consensus guidelines for advanced breast cancer (ABC3) capecitabine monotherapy is one of the recommended options even in first line (Cardoso et al, 2017).
  According to each center policy (minimum 1000 mg/m²) twice daily for 2 weeks followed by 1-week rest period, until progression or unacceptable toxicity
  Interventions: Drug: Capecitabine

INTERVENTIONS:
Drug: Darolutamide — treatment with darolutamide
  Arms: Arm 1 Darolutamide
Drug: Capecitabine — treatment with capecitabine
  Arms: Arm 2 Capecitabine

SUMMARY:
This is a multicenter uncontrolled, open-label, prospective, non-comparative randomized, phase II study. Patients will be randomized between darolutamide in Arm n°1 (two-stage Simon's design) and capecitabine in Arm n°2 with two patients randomized in Arm n°1 for one patient randomized in Arm n°2.

The trial population is composed of women over 18 years old with triple-negative and androgen receptor positive, locally recurrent (unresectable) or metastatic breast cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Woman, ≥18 years old;
2. Histologically confirmed locally recurrent (unresectable) or metastatic breast cancer;
3. Triple negative breast cancer:

   Estrogen receptor (ER)-negative and Progesterone receptor (PgR)-negative, as defined by a <10 % tumor stained cells by immunohistochemistry (IHC); HER2 negative status (i.e. IHC score 0 or 1+, or IHC score 2+ and FISH/SISH/CISH negative), confirmed centrally before inclusion with FFPE tissue from the primary tumour;
4. Androgen receptor (AR)-positive, as defined centrally by a ≥ 10% tumor stained cells by IHC Note: AR assessment by local pathologist before inclusion is not mandatory;
5. Patients with a relapse or progressive disease should be chemotherapy naïve or have received a maximum of one line of chemotherapy for advanced disease (providing they are not presenting with life-threatening metastasis); patients could have received adjuvant or neo-adjuvant therapy;
6. In the exceptional situation of pre-menopausal patient, the addition of a LHRH analog is recommended (androgens might act as an estrogen antagonist in premenopausal patients);
7. Presence of measurable or evaluable disease according to response evaluation criteria in solid tumors version 1.1 (RECIST v1.1)
8. Eastern cooperative oncology group (ECOG) ≤1;
9. Normal hematological function: Absolute neutrophile count (ANC) ≥1,500/mm³; platelets count ≥100,000/mm³; hemoglobin >10 g/dL; Note: subject must not have received any growth factor within 4 weeks or blood transfusion within 7 days of the hematology laboratory sample obtained at screening)
10. Normal hepatic function: total bilirubin ≤ 1.5 upper normal limit (UNL) unless this increase is due to a known Gilbert's disease; aspartate aminotransferase (ASAT) and alanine aminotransferase (ALAT) ≤2.5 UNL (or ≤5 UNL in case of hepatic metastasis);
11. Creatinine clearance (MDRD formula) ≥50 mL/min;
12. Systolic blood pressure (BP) <160 mm Hg and diastolic BP <95 mm Hg, as documented on day of registration/consent (Hypertension allowed provided it is currently controlled);
13. Cardiac ejection fraction ≥50% measured by multigated acquisition (MUGA) or echocardiography (ECHO) done within 4 weeks before inclusion;
14. For premenopausal patients, patient agreeing to use effective contraception during and for ≥6 months after completion of study treatment;
15. Patient able to comply with the protocol;
16. Patient must have signed a written informed consent form prior to any study specific procedures;
17. Patient must be affiliated to a Social Health Insurance.

Exclusion Criteria:

1. HER2-positive status (positivity defined as IHC3+ and/or FISH amplification ≥2);
2. Other concurrent malignancies, except adequately treated cone-biopsied in situ carcinoma of the cervix or basal cell or squamous cell carcinoma of the skin; patients who have undergone potentially curative therapy for a prior malignancy are eligible provided there is no evidence of disease for ≥5 years and patient is deemed to be at low risk for recurrence;
3. Active brain metastases or leptomeningeal disease; history of brain metastases allowed provided lesions are stable for at least 3 months as documented by head CT scan or Magnetic resonance Imaging (MRI) of the brain;
4. Non-malignant systemic disease, including active infection or concurrent serious illness that would make the patient a high medical risk;
5. Significant cardiovascular disease, including any of the following:

   1. NYHA class III-IV congestive heart failure
   2. Stroke, unstable angina pectoris or myocardial infarction within the past 6 months
   3. Severe valvular heart disease
   4. Ventricular arrhythmia requiring treatment;
6. Patients with rare hereditary problems of galactose intolerance, the Lapp lactase deficiency or glucose-galactose malabsorption should not be included;
7. Persistent toxicities grade ≥2 from any cause, except chemotherapy-induced alopecia and grade 2 peripheral neuropathy;
8. Any gastrointestinal disorder interfering with absorption of the study drug;
9. Difficulties with swallowing tablets;
10. An active viral hepatitis, known human immunodeficiency virus infection with detectable viral load, or chronic liver disease requiring treatment;
11. PREVIOUS TREATMENT IN THE METASTATIC SETTING: Previous treatment with: capecitabine (MET SETTING), first generation (bicalutamide) or second-generation AR inhibitors (enzalutamide, ARN-509, darolutamide) or other investigational AR inhibitors CYP17 enzyme inhibitor such as abiraterone (capecitabine in the adjuvant setting is allowed provided the last administration was at least ≥12 months prior to study entry)
12. Patients with known deficit of dihydropyrimidine dehydrogenase (DPD) activity; or in case of hypersensitivity to capecitabine or to any of its excipients or to fluorouracil;
13. Prior anticancer therapy within the last 3 weeks including radiotherapy, endocrine therapy, immunotherapy; chemotherapy (6 weeks for nitrosoureas and mitomycin C), or other investigational agents; concurrent palliative radiotherapy is allowed;
14. Concurrent enrolment in another clinical trial in which investigational therapies are administered;
15. Pregnant women, women who are likely to become pregnant or are breast-feeding;
16. Patients with any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule. Those conditions should be discussed with the patient before registration in the trial;
17. Patients with history of non-compliance to medical regimens or unwilling or unable to comply with the protocol;
18. Individual deprived of liberty or placed under the authority of a tutor.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — female
Enrollment: 94 (Actual)
Dates: Start 2018-03-14 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2022-07-20 (Actual)

PRIMARY OUTCOMES:
clinical benefit rate | at 16 weeks
  The clinical benefit rate (CBR) is the measurement of all patients who have a complete response (CR), partial response (PR) or stable disease (SD) at 16 weeks (CBR16) according to RECIST v1.1

SECONDARY OUTCOMES:
clinical benefit rate | at 24 weeks
  Clinical benefit rate (CBR24)
Objective response rate | at 16 and 24 weeks
  Objective response rate (ORR)
Duration of overall response | at 16 and 24 weeks
  Duration of overall response (DoR)
Overall survival | at 1 and 2 years
  Overall survival (OS)
Progression-free survival | at 1 and 2 years
  Progression-free survival (PFS)
Safety: Evaluation of toxicity in each arm according to CTCAE V4.03 | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  Evaluation of toxicity in each arm according to CTCAE V4.03

CONTACTS AND LOCATIONS:
Overall Officials: Hervé BONNEFOI, MD, Study Chair — Institut Bergonié - University of Bordeaux 2
Locations (1):
- Centre François Baclesse, Caen, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Bonnefoi H, Lerebours F, Pulido M, Arnedos M, Tredan O, Dalenc F, Guiu S, Teixeira L, Mollon D, Levy C, Verret B, Dawood H, Deiana L, Mouret Reynier MA, Augereau P, Canon JL, Huchet N, Guyonneau C, Lemonnier J, MacGrogan G, Goncalves A, Darbo E, Iggo R. Darolutamide or capecitabine in triple-negative, androgen receptor-positive, advanced breast cancer (UCBG 3-06 START): a multicentre, non-comparative, randomised, phase 2 trial. Lancet Oncol. 2025 Mar;26(3):355-366. doi: 10.1016/S1470-2045(24)00737-X. Epub 2025 Feb 17. PMID 39978376